CLINICAL TRIAL: NCT02632162
Title: Prevalence, Severity and Natural Course of Sleep Apnea After Cardiac Surgery
Acronym: SDB-ZRW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zürcher RehaZentrum Wald (Other)
Responsible Party: Sponsor
Other Study IDs: ZRW-SDB-2015
Record Dates: First submitted 2015-12-02; First posted 2015-12-16 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cardiac surgery: active Group screening
  Interventions: Other: screening
- orthopedic surgery: control Group screening
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — Screening for sleep disordered breathing with the ApnoeLink Air device

SUMMARY:
Sleep disordered breathing (SDB) is common in cardiovascular patients. Patients after cardiac surgery will be screened for SDB with the ApnoeLink device at the beginning of cardiac Rehabilitation and then after 3 weeks and 3 months.

DETAILED DESCRIPTION:
Objective(s) of the project

* Evaluate the prevalence of sleep apnea after cardiac surgery
* Compare results interindividually (group A vs. group B) and intraindividually (longitudinal assessment after 3 months)

Outcome(s)

* Prevalence of sleep apnoe at day 1 and 20 of rehabilitation and 3 months after cardiac surgery
* composite endpoint of events at 3 months (cardiovascular death, non-fatal myocardial infarction, non-fatal cardiac arrest, revascularisation procedure, new atrial fibrillation and stroke)
* change in 6-minute walking test (6-MWT)
* impact of heart surgery on sleep apnoe

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery or orthopedic surgery <2 weeks

Exclusion Criteria:

* known SDB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cardiac surgery < 2 weeks
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of SDB prevalence after cardiac surgery measured with ApnoeLink Air device | day 1, day 20, 3 months
  • Prevalence of sleep apnoe at day 1 and 20 of rehabilitation and 3 months after cardiac surgery assessed with the ApnoeLink Air device (ResMed)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hermann, MD, Principal Investigator — Zürcher RehaZentrum Wald
Locations (1):
- Zürcher RehaZentrum Wald, Wald, Switzerland